CLINICAL TRIAL: NCT07263841
Title: Comparison of Effectiveness of Tranexamic Acid Mesotherapy Versus Glutathione Mesotherapy in Post Burn Facial Hyperpigmentation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 435/RC/KEMU
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Post Burn Facial Hyperpigmentation
Keywords: hyperpigmentation; Mesotherapy; Effectiveness
MeSH Terms: conditions — Hyperpigmentation | interventions — Tranexamic Acid; Glutathione

STUDY DESIGN:
Intervention Model Description: each patient will be given both treatments, every participant will act as his own control.
Masking Description: outcome assessor will be masked to overcome biasness
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- fitzpatrick skin type3,4 patients of post burn facial hyperpigmentation will be included in this arm (Experimental): facial hyperpigmentation lesion will be divided into 2 halves and one treatment will be administered on each half
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — tranexamic acid decreases melanogenesis by inhibiting tyrosinase enzyme while glutathione converts eumelanin to pheomelanin
  Other Names: glutathione

SUMMARY:
INTERVENTION:

Patch test on forearm will be performed in all patients before starting treatment to check the sensitivity. Site of burn in the enrolled patients will include either cheek or forehead and total area (cm2) on each of above mentioned sites will be divided into two equal halves; one for tranexamic acid mesotherapy (maximum 5cm2) and other for glutathione mesotherapy (maximum 5cm2). Flip coin method will be used to decide which site and which half to be treated with tranexamic Acid or glutathione. Gentle cleansing of the affected area will be done Tranexamic acid is available in 500mg/5ml formulation, 1ml (100mg) of tranexamic acid will be taken and diluted in 10ml of 0.9% N/S i.e. 10mg/ml.This 10mg/ml of diluted formulation will be used for mesotherapy.

intradermally 1cm apart to the selected site using 1cc disposable syringe with 4mm depth 30G needle.4mm depth of intradermal injection will be controlled manually by the researcher on specific area of face. Maximum dose of tranexamic acid microinjections will not exceed 12.5 mg/5cm'.

Glutathione is available in 600mg powder formulation and will be prepared by dissolving in 5ml of distilled water. 1ml (120mg) of glutathione will be diluted in 10ml of 0.9% N/S i.e. 12mg/ml.This 12mg/ml of diluted formulation will be used for mesotherapy. Multiple microinjections, each 0.05ml (0.6mg) will be given intradermally 1cm apart to the selected site using 1cc disposable syringe with 4mm depth 30G needle. Maximum dose will not exceed 15mg/5cm2. All patients will be kept under observation for 20-30 minutes after each session to address any side effects (bruising, bleeding, pain etc.) and they will be advised to apply sunscreen of SPF 50 on whole of the face before sun exposure. After initial treatment session, patients will undergo six more treatment sessions with the same protocol at the interval of 2 weeks ( 2, 4, 6, 8, 10,12 weeks) and follow-up will be done monthly after the last session i.e. 4th, 5th and 6th month.

Final assessment will be done at 6th month. All clinical dermatoscopic photographs will be taken with Nikon D810 digital camera with dermlite 3 dermoscopy lens before the start of treatment, at each treatment session and then at each follow-up in same pre-settings, light and from same distance.

DETAILED DESCRIPTION:
Burn injuries are one of the leading cause of morbidity and mortality especially in developing countries. skin pigmentation disorders are one of the most frequent sequelae after burn injury while these conditions often improve over time,some are permanent and cause severe psychological disorders(specially on the face). 1 Inflammation of burnt skin triggers the melanocytes during the healing process which results in overproduction of melanin pigment that subsequently either gets dispersed to the epidermal keratinocytes or gets engulfed by the newly recruited macrophages leading to epidermal and dermal melanosis respectively. Unfortunately skin types with darker complexion due to melanosis (Fitzpatrick type III to IV), common in the subcontinent, are more susceptible to post inflammatory hyperpigmentation.1,2 A myriad of treatments including topical bleaching agents, chemical peels, tretinoins, sunscreens and various lasers have been used to prevent and reduce the hyperpigmentation with suboptimal results.

Tranexamic acid (TXA) is a novel agent used in the treatment of post burn hyperpigmentation, available in topical, oral and parentral formulations.3,4 The drug is widely used as anti-fibrinolytic agent and exerts its effects by inhibiting plasminogen-keratinocyte interaction leading to decrease in activity of tyrosinase enzyme thereby resulting in decrease synthesis of melanin from melanocytes.3,4 Human keratinocytes secrete plasminogen activator, which increases the plasmin production and melanogenesis.5 Blockade of this effect is the mechanism behind the therapeutic effect of tranexamic acid.6,7 Tranexamic acid mesotherapy can be a very good option for treating patients of post burn hyperpigmentation.

Glutathione (GSH) is widely used drug available in topical, oral and parenteral formulations with indications encompassing hyperpigmentation, anti-aging and antioxidant effects.8 It improves skin pigmentation by shifting melanogenesis from eumelanin (black brown in color) to pheomelanin (yellow red in color) through inhibiting tyrosinase enzyme, thus regulating the rate limiting step in melanin production.8,9 Glutathione is present intracellularly more abundantly in the reduced form (GSH) and is readily converted into its oxidized form (GSSG) in the process of scavenging free oxygen redicals and other toxins while trying to maintain the redox balance of cellular environment, as described by Sidarth sonthalia in his study. 9 Consequently the levels of glutathione are found to be decreased in the tissues experiencing metabolic stress due to various inflammatory processes like burns and other diseases i.e allergies, melasma and malignancies. 8,9 In our study, we will use mesotherapy, which is an effective way of delivering de-pigmentation drugs like tranexamic acid and glutathione directly into the dermis which is the nidus of ongoing inflammatory process in the burn wounds while avoiding the undesirable consequences of systemic therapy.7,10 There is limited data about the regimen protocol and quantitative comparison of these two types of mesotherapies. This will be the first study on local and international level for measurement of post burn facial hyperpigmentation as to date there are no reliable objective methods for measuring skin hyperpigmentation quantitatively in this population of patients. Our study, with availability of ideal population sample from one of the largest burn centre in the country, will surely add to scarce knowledge currently published in literature regarding the use of tranexamic acid and glutathione to overcome hyperpigmentation. This can lower the psychosocial stigmata of post burn marks and ease the way of burn survivors for re-integration into society.

6.4 OBJECTIVE:

To compare the quantitative effectiveness of tranexamic acid mesotherapy versus glutathione mesotherapy in post burn facial hyperpigmentation.

6.5 OPERATIONAL DEFINITIONS: Post burn facial hyperpigmentation It is the condition of facial skin in which there is pigmentation of skin that follows the burn injuries i.e self-healed burns managed conservatively without skin grafting.

Mesotherapy Mesotherapy is a procedure in which multiple microinjections of tranexamic acid or glutathione will be given 1 cm apart for treating post burn facial hyperpigmentation.

Effectiveness

Effectiveness is the reduction in hyperpigmentation at 6 month follow-up and will be measured objectively as skin hyperpigmentation index (SHI) score using online digital processing system and SHI score ≤2 will be considered effective and graded as:

0-1 excellent responce 1-2 moderate response 2-3 mild response 3-4 no responce 6.6 HYPOTHESIS Tranexamic acid mesotherapy is more effective as compared to glutathione mesotherapy for reduction of pigmentation in post burn facial hyperpigmentation patients.

6.7 MATERIAL AND METHODS Study Design Randomized control trial. Setting Outpatient Department of Plastic surgery, King Edward medical University/ Mayo Hospital, Lahore.

Duration of Study Study will be completed within 6 months after approval of synopsis. Sample size Sample size of 60 patients is estimated by using 5% level of significance, 90% power of test with expected %age efficacy of tranexamic acid as 79% and of glutathione as 37.5% 10

* Level of significance = 5% 1-β=Power of test 90% P1=%age excellent response with TA = 78% P2=%age excellent response with Glutathione = 37.5% n =60

Sampling Technique Non-probability convenient sampling

SELECTION CRITERIA:

Inclusion Criteria Both sexes of WHO adult age group 18-65 years . Patients with healed facial burns managed conservatively without skin grafting.

From 6 month to 12 month post burn injury (patient enrollment to be done before scar maturation starts) Patients with Fitzpatrick skin types III to IV. Patients with mental capacity to give informed consent. Exclusion Criteria Patients with documented hypersensitivity reactions to either drug or dressing etc.

History of de-pigmentation treatment, phototherapy. Healed burn wounds with hypertrophic scar. History of bleeding or clotting disorders, renal disease, collagen vascular disease and other photodermatoses3.

Pregnant or lactating females3. Patients on hormone replacement therapy, oral contraceptives, concomitant use of anticoagulant, or any photosensitizing drug3.

6.8 DATA COLLECTION PROCEDURE: Data will be collected using a pre-designed preform. Sixty patients (Fitzpatrick skin type III to IV) will be enrolled in this study. Patient's demographics and skin type will be noted. Written informed consent will be taken from the patients fulfilling the inclusion criteria from outpatient department of KEMU/ Mayo Hospital, Lahore.

PATIENT ASSESSMENT Patient will be assessed clinically at 2 weeks intervals using Skin hyperpigmentation index (SHI), which is a fully automated and standardized method for the quantitative assessment of skin pigmentation. Clinical photographs of pigmented and normal sun-protected unexposed area of body from same patient (L4 spinous process as reference point) will be uploaded in software to calculate skin hyperpigmentation index using following formula10 .

PSArea with hyperpigmentation SHI= __________________________ PSReference point

PS =skin pigmentation

SHI score will be graded as:

0-1= No hyperpigmentation: Excellent response 1-2= Light hyperpigmentation: Moderate response 2-3= Medium hyperpigmentation: Mild response 3-4= Severe hyperpigmentation: No response

.

6.9 DATA ANALYSIS PROCEDURE: Data will be entered and analyzed by using SPSS 26 (IBM SPSS statistics for windows, version 26.0 NY: IBM corp). Quantitative variables like SHI score will be presented as mean and standard deviation. Qualitative variables like gender will be presented as frequency and percentages and analysed by chi-square. For Comparison of effectiveness of tranexamic acid mesotherapy and glutathione mesotherapy we will apply sample t-test if normally distributed. P value <0.05 will be considered significant.

6.10 OUTCOME & UTILIZATION: Post burn facial hyperpigmentation is a very common problem especially in women. Its management is challenging because it runs a chronic course producing significant emotional and psychological effects in patients. There is limited efficacy of oral and local treatments and they require prolonged usage which leads to disappointment in patients. So, we have designed a study in which tranexamic acid mesotherapy and glutathione mesotherapy will be done in such patients and effectiveness of both will be compared quantitatively. Also, it will be the first study in Pakistan on quantitative comparison of tranexamic acid and glutathione mesotherapy in post burn hyperpigmentation. Perhaps in the near future, one of the studied options will be considered potentially efficacious and safe in the treatment of post burn facial hyperpigmentation. This will help to implement a better management of facial hyperpigmentation in burn patients to improve their quality of life and social integration.

ELIGIBILITY:
Inclusion Criteria:● Both sexes of WHO adult age group 18-65 years .

* Patients with healed facial burns managed conservatively without skin grafting.
* From 6 month to 12 month post burn injury (patient enrollment to be done before scar maturation starts)
* Patients with Fitzpatrick skin types III to IV.
* Patients with mental capacity to give informed consent.

Exclusion Criteria:● Patients with documented hypersensitivity reactions to either drug or dressing etc.

* History of de-pigmentation treatment, phototherapy.
* Healed burn wounds with hypertrophic scar.
* History of bleeding or clotting disorders, renal disease, collagen vascular disease and other photodermatoses3.
* Pregnant or lactating females3.
* Patients on hormone replacement therapy, oral contraceptives, concomitant use of anticoagulant, or any photosensitizing drug3.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-26 (Estimated); Study Completion 2026-03-26 (Estimated)

PRIMARY OUTCOMES:
improvement in facial hyperpigmentation | 6months
  patients will be assessed for improvement in hyperpigmentation by skin hyperpigmentation index till 6 months after completion of sessions

CONTACTS AND LOCATIONS:
Overall Officials: Assistant Professor Plastic surgery, MBBS, FCPS Plastic Surgery, MD, Study Director — Mayo Hospital,KEMU,Lahore
Locations (1):
- King Edward Medical University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
privacy concerns of patient

REFERENCES:
- [Background] Isseroff RR, Rifkin DB. Plasminogen is present in the basal layer of the epidermis. J Invest Dermatol. 1983 Apr;80(4):297-9. doi: 10.1111/1523-1747.ep12534677. PMID 6339645